CLINICAL TRIAL: NCT04546165
Title: Efficacy of Manual Therapy in Tension-type Headache Patients With Neck Pain: A Randomized Controlled Trial
Brief Title: Manual Therapy in Tension-type Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Mustafa Corum, Principal Investigator, Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020/289
Record Dates: First submitted 2020-09-06; First posted 2020-09-11 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Tension-Type Headache
MeSH Terms: conditions — Tension-Type Headache | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- manipulation group (Active Comparator): manipulation plus exercise
  Interventions: Procedure: suboccipital inhibition plus exercise; Procedure: exercise
- myofascial release group (Active Comparator): suboccipital inhibition plus exercise
  Interventions: Procedure: manipulation plus exercise; Procedure: exercise
- exercise group (Active Comparator): only exercise
  Interventions: Procedure: manipulation plus exercise; Procedure: suboccipital inhibition plus exercise

INTERVENTIONS:
Procedure: manipulation plus exercise — HLVA manipulation was performed for 8 sessions (twice a week for four weeks) using a segment-specific technique for segmental dysfunctions of the upper cervical spine. . By bringing the cervical spine to light flexion and about 15-20º lateral flexion without any rotational motion, the middle finger of the manipulating hand provided deep contact, and an HVLA thrust was applied out of the rotational slack by applying a deep force from the dorsal to the ventral direction
  Arms: exercise group; myofascial release group
Procedure: suboccipital inhibition plus exercise — Suboccipital inhibition was performed for 8 sessions (twice a week for four weeks) as a combined muscle and soft tissue inhibition technique. While the patient was in the supine position, the physician sitting at the top end of the table placed the fingers of both hands on the patient's suboccipital region
  Arms: exercise group; manipulation group
Procedure: exercise — Patients were asked to exercise at least three days a week during treatment. The exercise program, which lasted 20 to 30 minutes, included cervical range of motion (ROM) exercises to warm-up and cool-down, and then stretching exercises of cervical and upper thoracic spine muscles (trapezius, levator scapula, sternocleidomastoid) and strengthening exercises (cervical isometric contraction and concentric contraction of the deep cervical flexor muscles).
  Arms: manipulation group; myofascial release group

SUMMARY:
Tension-type headache (TTH) causes a significant negative impact on working and daily life due to the reduction in work productivity and family and social activities causes. There is evidence that manual therapy and exercise reduce nociceptive input from the cervical spine and surrounding muscles, the use of manual therapy in TTH management

DETAILED DESCRIPTION:
Increased cranio-cervical muscle sensitivity is the most prominent finding in TTH. Also, neck pain is markedly more common in individuals with TTH compared with the control population (88.4%, and 56.7%, respectively). Therefore, current research on the pathogenesis of TTH focuses on the role of musculoskeletal disorders in the cervical spine and the facilitation of nociceptive pain processing. It has been suggested that peripheral sensitivity of nociceptors in cranio-cervical muscles and other cervical structures, as well as sensitivity of nociceptive pain pathways in the central nervous system (CNS) due to long-term nociceptive stimuli may play a role in development and chronification of TTH

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of TTH was made based on the International Classification of Headache Disorders criteria, third edition (ICHD-3 beta)
* (bilateral localization, pressing and tightening pain, mild-moderate intensity [≤7.0 on a visual analog scale (VAS)]
* no increase in pain during physical activity
* patients did not report any photophobia, phonophobia, vomiting or nausea, as requested by the ICHD-III diagnostic criteria
* had symptoms for more than 3 months
* the patients had to have had at least one segmental dysfunction of the upper cervical spine in all groups (by functional and pain-provocation tests).

Exclusion Criteria:

* any other primary or secondary headache according to the ICHD-III criteria
* a history of neck or head trauma (e.g., whiplash)
* any red flags (vertebral tumor, fracture, dislocation and infection, metabolic diseases, rheumatic and connective tissue diseases, systemic neuromuscular diseases, prolonged history of steroid use)
* diagnosis of any structural spinal disorders (osteoporosis, disc herniation, myelopathy, spinal stenosis, spondylolisthesis)
* prior surgery to the cervical spine
* application of other treatment methods such as physical therapy or anesthetic block to the head and neck area within the last 3 months
* initiation of pharmacologic prophylaxis within two months prior to randomization
* pregnancy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2020-06-22 (Actual); Primary Completion 2020-09-10 (Actual); Study Completion 2020-09-10 (Actual)

PRIMARY OUTCOMES:
Headache Frequency (HF) | Changes from baseline in Headache Frequency Score to 1 month and 3 months
  . Headache frequency was measured as the total number of days with headache (days/2-week) in the previous 2 weeks.

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) | Changes from baseline in Visual Analog Scale Score to 1 month and 3 months
  The self-evaluation of pain severity of headache and neck pain during rest and activity in the previous week was calculated using a 10-cm VAS scale, where 0 in the left corner of the scale represented 'no pain' and 10 in the right corner represented 'the worst pain that could be imagined'
Headache Impact Test-6 (HIT-6) | Changes from baseline in Headache Impact Test-6 Score to 1 month and 3 months
  The total score was calculated in HIT-6, which consisted of 6 questions with 5 answer options for each (never: 6 points, rarely: 8 points, sometimes: 10 points, very often: 11 points, always: 13 points). A total score of 36 means best and 78 means worst in terms of headache
Neck Disability Index (NDI) | Changes from baseline in Neck Disability Index Score to 1 month and 3 months
  The NDI consists of 10 questions about pain disability in the neck region ("no disability" = 0, and "full disability" = 5). The total NDI score was calculated, with 0 showing the best score and 50 showing the worst score.
Pressure-Pain Threshold (PTT) | Changes from baseline in Pressure-Pain Threshold Score to 1 month and 3 months
  PPT measurements were performed using a mechanical pressure algometer on the temporalis anterior muscle The feeling of pressure was gradually increased until it turned into pain or discomfort, at which point the pressure value was recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Corum, MD, Study Chair — Istanbul Physical Medicine Rehabilitation Training & Research Hospital
Locations (1):
- Istanbul Physical Medicine and Rehabilitation Training and Research Hospital, Istanbul, Bahcelievler, Turkey (Türkiye)